CLINICAL TRIAL: NCT06578260
Title: Support Groups - a Model for Social Inclusion and Reduction of Bullying in School
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Lisbeth Valla, Associate Professor Lisbeth Valla, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 717417
Record Dates: First submitted 2024-08-16; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Bullying
Keywords: Supportgroups; schoolchildren; solution-focused-approach
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled trial (CRCT)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect and outcomes in the intervention schools (Experimental): The intervention schools will use the Support Group intervention regarding bullying and exclusion.
  Interventions: Behavioral: Peer support groups with a solution-focused approach
- The outcomes in the control schools (No Intervention): The control schools will implement the same measures as they normally do regarding bullying and exclusion.

INTERVENTIONS:
Behavioral: Peer support groups with a solution-focused approach — To investigate the effectiveness of a support group intervention using a solution-focused approach among school children in 5th-7th grade in southeastern Norway
  Arms: The effect and outcomes in the intervention schools

SUMMARY:
Study Title: Support Groups - a model for social inclusion and reduction of bullying in school Study Design: Cluster Randomized Controlled trial (CRCT) Objective: To investigate the effectiveness of a support group intervention using a solution-focused approach among school children in 5th-7th grade in southeastern Norway Intervention: Peer support groups with a solution-focused approach Study Population: School Children

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the effectiveness of a support group intervention using a solution-focused approach in reducing bullying, enhancing mental health, improving quality of life, and increasing general self-efficacy among school children in 5th-7th grade. Investigators hypothesize that the awareness of bullying created by the intervention, and the empowerment of children as contributors to the solution, will generate positive ripple effects benefiting all children in the intervention schools. Furthermore, investigators hypothesize that children with a peer support group will exhibit lower levels of bullying, improved mental health, better quality of life, and increased general self-efficacy after the intervention compared to their baseline levels. Investigators expect these effects to persist even after 3 and 6 months. Aligned with the cluster RCT, the investigators will undertake a parallel process evaluation to assess the extent of the intervention coverage, whether the intervention was implemented according to the protocol, and identify factors that hinder or aid the implementation of a support group intervention. For the process evaluation, investigators will use the framework presented by the Medical Research Council guidelines focusing on the implementation (what is implemented and how), the mechanisms of impact (how the delivered intervention produces change), and the context (how the context affects implementation and outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Primary Schools with more than 200 students
* Public Health Nurse employed in a 50% position or more

Exclusion Criteria:

* Primary Schools with less than 200 students

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1586 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Bullying- change from baseline in bullying using the Olweus questionnaire at end of intervention, 3 months and 6 months after end of intervention on individual level at intervention schools. | Baseline, Week 6, Week 18 and Week 32
  The Olweus questionnaire is a validated self-reported questionnaire that may be answered from ; Not at all (no bullying), one or seldom, 2-3 times in the months or about one times a week or more (worst possible bullying score) (Olweus, 2013).
Mental health- change from baseline in mental health using the Strength and Difficulties Questionnaires (SDQ), at end of intervention, 3 months and 6 months after end of intervention on individual level at intervention schools. | Baseline, Week 6, Week 18 and Week 32
  The Strength and Difficulties Questionnaires (SDQ) is a validated self-reported questionnaire which consists of 25-items (Goodman, 1999).
  The questionnaires measure emotional problems, conduct problems, hyperactivity, peer problems, pro-social behavior and impact score. The questionnaires may be answered form "not true" (lowest possible score) to "certainly true" (highest possible score). A high total difficulties score indicates that the individual is experiencing a high level of difficulties, while a low score indicates a low level of difficulties.
Self-efficacy-change from baseline in self-efficacy using the General self-efficacy scale, at end of intervention, 3 months and 6 months after end of intervention on individual level at intervention schools. | Baseline, Week 6, Week 18 and Week 32
  The General self-efficacy scale is a self-administered form with five response categories from "Completely agrees to "not agrees". The scale measures the belief in self-efficacy. Highest scores indicate best self-efficacy (Bandura, 1997).
Quality of life-change from baseline in quality of life using the Kidscreen -10, 4 months after baseline, end of intervention and 6 months after end of intervention in both intervention and control schools in 5th to 7th grade on class level. | Baseline, Week 17, Week 30 and Week 56
  The KIDSCREEN-10 index is the shortest version of the KIDSCREEN questionnaires and measures general health-related quality of life (Detmar, Bruil, Ravens-Sieberer, Gosch & Bisegger, 2006). Possible scores range from "not at all" or "never" (lowest possible score) to "a high degree" or "always" (highest possible score).
Class environment- change from baseline using the Norwegian student survey (Elevundersøkelsen), 4 months, end of intervention and 6 months after end of intervention in both intervention and control schools in 5th to 7th grade on class level. | Baseline, Week 17, Week 30 and Week 56
  To measure class environment all children in 5th to 7th grade will complete the Norwegian student survey (Elevundersøkelsen, UDIR 2023). The survey which asking among other things about bullying and inclusion in the school environment and peer relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Valla, Phd, Principal Investigator — OsloMet
Locations (1):
- OsloMet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06578260/Prot_000.pdf
  • Informed Consent Form (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06578260/ICF_001.pdf